CLINICAL TRIAL: NCT01217411
Title: Two Phase I Studies in Patients With Brain Metastases From Any Primary Histology, Followed by a Randomized Phase 2 Study of RO4929097 Combined With CNS Radiotherapy in Patients With Brain Metastases From Breast Cancer Whose Tumors Are Estrogen Receptor Negative
Brief Title: RO4929097 and Whole-Brain Radiation Therapy or Stereotactic Radiosurgery in Treating Patients With Brain Metastases From Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Other - Protocol moved to Administratively Complete
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02533; NCI-2011-02533 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000686136; MDA-2009-0582; 2009-0582 (Other: M D Anderson Cancer Center); 8543 (Other: CTEP); N01CM00039 (NIH); P30CA016672 (NIH); U01CA062461 (NIH); U01CA069852 (NIH); U01CA076576 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2015-02-06 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Adult Solid Neoplasm; Extensive Stage Lung Small Cell Carcinoma; HER2/Neu Negative; HER2/Neu Positive; Male Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Recurrent Breast Carcinoma; Recurrent Lung Non-Small Cell Carcinoma; Recurrent Lung Small Cell Carcinoma; Recurrent Melanoma; Stage IV Breast Cancer AJCC v6 and v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Breast Neoplasms, Male; Brain Neoplasms; Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Melanoma | interventions — Mental Status and Dementia Tests; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Radiosurgery

ARMS (2):
- Arm I (WBRT or SRS) (Active Comparator): Patients with >= 4 brain lesions undergo WBRT as in phase I and patients with =< 3 brain lesions undergo SRS as in phase I.
  Interventions: Procedure: Cognitive Assessment; Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Radiosurgery; Radiation: Whole-Brain Radiotherapy
- Arm II (WBRT or SRS and RO4929097) (Experimental): Patients with >= 4 brain lesions receive RO4929097 and undergo WBRT as in phase I and patients with =< 3 brain lesions receive RO4929097 and undergo SRS as in phase I.
  Interventions: Procedure: Cognitive Assessment; Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Radiation: Stereotactic Radiosurgery; Radiation: Whole-Brain Radiotherapy

INTERVENTIONS:
Procedure: Cognitive Assessment — Ancillary studies
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: R04929097; RG-4733; RO4929097
  Arms: Arm II (WBRT or SRS and RO4929097)
Other: Laboratory Biomarker Analysis — Correlative studies
Radiation: Stereotactic Radiosurgery — Undergo SRS
  Other Names: SRS; Stereotactic External Beam Irradiation; stereotactic external-beam radiation therapy; Stereotactic Radiation Therapy; Stereotactic Radiotherapy; stereotaxic radiation therapy; stereotaxic radiosurgery
Radiation: Whole-Brain Radiotherapy — Undergo WBRT
  Other Names: WBRT; whole-brain radiation therapy

SUMMARY:
This randomized phase I/II trial studies the side effects and the best dose of RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097) when given together with whole-brain radiation therapy or stereotactic radiosurgery and to see how well it works compared to whole-brain radiation therapy or stereotactic radiosurgery alone in treating patients with breast cancer or other cancers (such as lung cancer or melanoma) that have spread to the brain. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Whole-brain radiation therapy uses high energy x-rays deliver radiation to the entire brain to treat tumors that can and cannot be seen. Stereotactic radiosurgery may be able to deliver x-rays directly to the tumor and cause less damage to normal tissue. It is not yet known whether giving RO4929097 together with whole-brain radiation therapy or stereotactic radiosurgery may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum-tolerated dose (MTD) and phase II dose of RO4929097 when combined with whole-brain radiation therapy (WBRT). (Phase I) II. Determine the safety profile of RO4929097 when combined with WBRT. (Phase I) III. Determine the MTD and phase II dose of RO4929097 when combined with stereotactic radiosurgery (SRS). (Phase I) IV. Determine the safety profile of RO4929097 when combined with SRS. (Phase I) V. Determine whether the addition of RO4929097 to WBRT or SRS significantly increases the percentages of estrogen receptor-negative breast cancer patients with brain metastases who achieve response (complete response [CR] + partial response [PR]) in the brain at the 12-week (3-month) time point after cranial radiotherapy. (Phase II)

SECONDARY OBJECTIVES:

I. Correlate responses and time to progression to: pre- and post-therapy tumor and archived tumor tissue expression of molecular and stem cell markers; pre- and post-therapy plasma biomarkers; changes in pre- and post-therapy tumor and archived tumor tissue expression of molecular and stem cell markers over the first 5 days of therapy and changes of pre- and post-therapy plasma biomarkers over the course of therapy; in Notch positive and Notch negative tumors, over the first 5 days of therapy with RO4929097, compare tumor tissue expression of molecular and stem cell markers. (Phase I and II) II. Determine progression free survival (PFS) in the brain for each treatment arm. (Phase II) III. Determine the percentage of patients alive and disease free (in the brain) at 6 months. (Phase II) IV. Determine local control rate (in the brain) at 24- and 48-week time point after cranial radiotherapy for each treatment arm. (Phase II) V. Determine distant failure rate (in the brain) at 24- and 48-week time point after cranial radiotherapy for each treatment arm. (Phase II) VI. Determine PFS in the body for each treatment arm. (Phase II) VII. Determine systemic response rate. (Phase II) VIII. Determine percentage of patients alive and without progression systemically at 6 months. (Phase II) IX. Further describe the safety profile of each treatment arm. (Phase II) X. Compare neurocognitive outcomes in each treatment arm. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of gamma-secretase/Notch signalling pathway inhibitor RO4929097 followed by a randomized phase II study.

PHASE I: Patients with >= 4 brain lesions receive RO4929097 orally (PO) once daily (QD) on days 1-3 weekly beginning 1 day prior to the first day of WBRT and continuing for 6 weeks (42 days) after the completion of radiation therapy. Patients with >= 4 brain lesions also undergo whole-brain radiotherapy (WBRT) once daily, 5 days a week, for 2-4 weeks beginning on day 2. Patients with =< 3 brain lesions receive RO4929097 PO QD on days 1-7 in weeks 1 and 2 and then days 1-3 in all subsequent weeks beginning 2 days prior to the first day of SRS and continuing for 6 weeks (42 days) after the completion of radiation therapy. Patients with =< 3 brain lesions also undergo stereotactic radiosurgery (SRS) on day 4. Treatment continues in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients with >= 4 brain lesions undergo WBRT as in phase I and patients with =< 3 brain lesions undergo SRS as in phase I.

ARM II: Patients with >= 4 brain lesions receive RO4929097 and undergo WBRT as in phase I and patients with =< 3 brain lesions receive RO4929097 and undergo SRS as in phase I.

After completion of study treatment, patients are followed up every 12 weeks for up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have histologically or cytologically confirmed breast cancer or other cancers (such as lung cancer, melanoma, etc) with newly diagnosed metastatic disease to the brain will be eligible for the Phase 1 study only, however, those patients who have available systemic therapeutic options with a demonstrated survival benefit will not be eligible; for Phase 2, patients must have histologically or cytologically confirmed estrogen receptor negative breast cancer with newly diagnosed metastatic disease to the brain
* Patients must have measurable disease in the brain, defined as at least one lesion that can be accurately measured in at least two dimensions (longest diameter and its longest perpendicular diameter to be recorded)
* There is no limit on type or number of prior therapies, except that prior therapy with notch inhibitors is not allowed, and patients should not have received prior cranial radiation; therapy naïve patients are eligible; at least 14 days (2 weeks) must have elapsed from any prior experimental therapy, chemotherapy or radiotherapy; toxicities from prior chemotherapy or radiotherapy should have resolved to < grade 2; patients with newly diagnosed brain metastases who have received therapeutic regimens with well-characterized, delayed toxicity (e.g. hematologic toxicity observed following carmustine [BCNU] or mitomycin C) will not receive experimental therapy until the patient has adequately recovered from all drug related toxicities
* Karnofsky performance status (KPS) >= 70%; Recursive Partitioning Analysis (RPA) class I or II; a small feasibility cohort of 10 RPA class III (KPS < 70%) patients may be enrolled, however these patients, if enrolled will not be included in the efficacy analysis
* Hemoglobin >= 9g/dL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limits of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Tumor HER2/neu status may be positive or negative
* Women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately; prior to dispensing RO4929097, the investigator must confirm and document the patient's agreement to the use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
* Ability to understand and the willingness to sign a written informed consent document
* A tumor site (outside the central nervous system) for needle biopsy for research purposes is preferable
* Ability to swallow pills

Exclusion Criteria:

* At least 14 days (2 weeks) must have elapsed from any prior experimental therapy, chemotherapy or radiotherapy; toxicities from prior chemotherapy or radiotherapy should have resolved to < grade 2
* Patients may not be receiving any other investigational agents
* Patients with leptomeningeal metastases should be excluded from this clinical trial
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Patients taking medications that are generally accepted by the QTdrugs.org Advisory Board to carry a risk of torsades de pointes, including antiemetics, are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP450 family 3, subfamily A, polypeptide 4 (CYP3A4) and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; if such patients cannot be switched to alternative medications, they will be ineligible to participate in this study
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption; patients must be able to swallow tablets
* Patients who are known to be serologically positive for hepatitis A, B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, and hypokalemia; uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV), unstable angina pectoris, a history of torsades de pointes or other significant cardiac arrhythmias, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with RO4929097
* Cardiovascular: baseline QTcF > 450 msec (male) or QTcF > 470 msec (female)
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are not eligible to participate in this study
* A requirement for antiarrhythmics or other medications known to prolong QTc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-10-01 (Actual); Primary Completion 2011-11-30 (Actual); Study Completion 2011-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Groves, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - M D Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 1, 2010 to December 21, 2011. All recruitment was done in a medical clinic setting.
Pre-assignment Details: Study terminated early due to low accrual and discontinuation of investigational study drug.
Groups:
- Phase 1 Arm I (WBRT + R04929097): Patients with >= 4 brain lesions undergo WBRT + R04929097
  Whole-brain radiation therapy (WBRT): Undergo radiotherapy; 30-40 Gy over 10-20 fractions for patients with 4 or more brain lesions, or who are otherwise not eligible or appropriate for stereotactic radiosurgery
- Phase 1 Arm II (SRS + RO4929097): Patients with =< 3 brain lesions receive RO4929097 and undergo SRS. For the SRS regiment: RO4929097 on Days 1-7 (no drug on days 8-14), weeks 1 and 2 only.
  Stereotactic radiosurgery (SRS): Undergo radiosurgery; 20 Gy for tumors up to 1cm diameter, 18 Gy for tumors from 1.1-2.5 cm, 16 Gy for tumors >2.5 cm for patients with 3 or fewer brain lesions, and if overall patient status and tumor geometry amenable to this treatment modality
Period: Overall Study
Arm/Group | Phase 1 Arm I (WBRT + R04929097) | Phase 1 Arm II (SRS + RO4929097)
Started | 3 | 2
5mg | 3 | 2
10mg | 0 | 0
20mg | 0 | 0
Completed | 0 | 0
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: 5 participants were enrolled/treated at the 5 mg (starting dose) study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Arm I (WBRT + R04929097) | Phase 1 Arm II (SRS + RO4929097) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Continuous [Median (Full Range); unit: years] | 49 [30 to 56] | 49 [30 to 56] | 49 [30 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 Arm I Maximum-tolerated Dose (MTD) of RO4929097 in Combination With Whole-brain Radiotherapy (WBRT)
Description: Maximum-tolerated dose (MTD) of RO4929097 in combination with WBRT, determined according to incidence of dose limiting toxicity (DLT) graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I)
Time Frame: 4 weeks
Population: Analysis was not available due to small number of patients on the study.
Groups:
- Phase 1 Arm I: RO4929097 dose to be determined; Dosing cohorts: 5 mg, 10 mg and 20 mg
  For patients with 4 or more lesions: Phase I WBRT+RO4929097; Begin RO4929097** (3 days on/4 days off continuous) 1 day prior to beginning WBRT
Arm/Group | Phase 1 Arm I
Number analyzed (Participants) | 0

2. Primary Outcome: Phase 1 Arm II MTD of RO4929097 in Combination With Stereotactic Surgery (SRS)
Description: MTD of RO4929097 in combination with SRS, determined according to incidence of DLT graded using the NCI CTCAE version 4.0 (phase I)
Time Frame: 4 weeks
Population: Analysis was not available due to small number of patients on the study.
Groups:
- Phase I Arm II: RO4929097 dose to be determined; Dosing cohorts: 5 mg, 10 mg and 20 mg
  For patients with 3 or fewer lesions: Phase I SRS + RO4929097; Begin RO4929097** (3 days on/ 4 days off continuous) 2 days prior to SRS
Arm/Group | Phase I Arm II
Number analyzed (Participants) | 0

3. Primary Outcome: Response Rate (Complete or Partial Response)
Description: Only participants with measurable disease present at baseline, received at least 6 weeks of therapy, and had disease re-evaluated considered evaluable for response. Complete Response (CR): Disappearance all lesions; Partial Response (PR): =/>50% decrease in sum bidimensional products all lesions reference baseline sum of bidimensional products of all lesions; Progressive Disease (PD): >25% increase in sum bidimensional products of lesions, or progression of any treated lesion not target lesion, or appearance of 1 or > new lesions at least 6 mm in unidimensional size. Stable Disease (SD): Neither sufficient shrinkage for PR nor increase for PD, reference smallest sum of bidimensional products of all lesions.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Phase I Arm I: Arm 1: Patients with 4 or more lesions will receive Whole Brain Radiation Therapy (WBRT) combined with R04929097 (study drug) 1st cohort: Starting dose of 5mg (2nd cohort 10mg, 3rd cohort 20mg) (3 days on/4 days off continuous) 1 day prior to beginning WBRT
- Phase 1 Arm II: Arm 2: Patients with less than 4 lesions will receive Stereotactic Radiosurgery (SRS) combined with R04929097 (study drug). 1st cohort: starting dose of 5mg (2nd cohort 10mg, 3rd cohort 20 mg) (3 days on/4 days off continuous) 3 days prior to SRS)
Arm/Group | Phase I Arm I | Phase 1 Arm II
Number analyzed (Participants) | 3 | 2
Participants | 3 | 2

ADVERSE EVENTS:
Time Frame: Routine adverse event (AE) monitoring and reporting till 30 days following the last dose of the Investigational Agent, up to 16 weeks total.
Description: Study did not progress to Phase II so two arms of second phase excluded from AE reporting table.
Groups:
- Phase 1 Arm I (WBRT + R04929097): RO4929097 dose to be determined; Dosing cohorts: 5 mg, 10 mg and 20 mg
  For patients with 4 or more lesions: Phase I WBRT+RO4929097; Begin RO4929097** (3 days on/4 days off continuous) 1 day prior to beginning WBRT
  For patients with 3 or fewer lesions: Phase I SRS + RO4929097; Begin RO4929097** (3 days on/ 4 days off continuous) 2 days prior to SRS
Arm/Group | Phase 1 Arm I (WBRT + R04929097) | Phase 1 Arm II (SRS + RO4929097)
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Arm I (WBRT + R04929097) (N=3) | Phase 1 Arm II (SRS + RO4929097) (N=2)
Anemia (Cardiac disorders) | 1 (1) | 0
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0
Death NOS (General disorders) | 1 (1) | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Arm I (WBRT + R04929097) (N=3) | Phase 1 Arm II (SRS + RO4929097) (N=2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0
Anemia (Blood and lymphatic system disorders) | 2 (4) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Cardiac disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (4) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4) | 1 (5)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (5) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Investigations (Investigations) | 3 (9) | 2 (8) — Increased: Phosphorus, Protein, Albumin, Co^2, Chloride Serum Elevated Lactate Dehydrogenase (LDH); Decreased: Creatinine Kinase, Chloride Serum, Decreased aspartate aminotransferase (AST) (AST/SGOT), Chloride Serum, and Uric Acid
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle Wasting (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Syncope (Psychiatric disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Darkness skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to small number of patients enrolled on study, researchers were unable to make meaningful conclusions from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less